CLINICAL TRIAL: NCT04218708
Title: Electronic Cigarettes as a Harm Reduction Strategy Among People Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01179
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Nicotine Addiction
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Chewing Gum; Insemination, Artificial, Heterologous; Ethanol; Smoking Devices; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- counseling + nicotine replacement therapies NRT (Active Comparator): A research assistant (RA) trained in motivational interviewing and qualitative methods will support the PI to deliver counseling sessions and conduct interviews. Briefly, during each visit, with help of the RA, participants will provide exhaled CO and saliva cotinine test, and complete surveys in REDCAP using a tablet, allowing programmed logic checks and skip patterns to minimize burden. The RA will also deliver brief motivational counseling tailored to the participant's readiness to quit and arm in the study (NRT). Participants will also receive their NRT to last them to the following visit based on their baseline smoking.
  Interventions: Other: Nicotine patch and gum; Behavioral: Minnesota Nicotine Withdrawal Scale (MNWS); Behavioral: ASSIST (the Alcohol, Smoking and Substance Involvement Screening); Behavioral: Counseling
- Counseling + Standardized Research E-cigarettes (SREC) (Active Comparator): Participants in the SREC arm to practice using the SREC and give them instructions to return with their SREC and used refill tanks on every visit. A research assistant (RA) trained in motivational interviewing and qualitative methods will support the PI to deliver counseling sessions and conduct interviews. Briefly, during each visit, with help of the RA, participants will provide exhaled CO and saliva cotinine test, and complete surveys in REDCAP using a tablet, allowing programmed logic checks and skip patterns to minimize burden. The RA will also deliver brief motivational counseling tailored to the participant's readiness to quit and arm in the study (SREC). Participants will also receive their SREC to last them to the following visit based on their baseline smoking.
  Interventions: Behavioral: Minnesota Nicotine Withdrawal Scale (MNWS); Behavioral: ASSIST (the Alcohol, Smoking and Substance Involvement Screening); Behavioral: Counseling; Other: NIDA Standardized Research E-cigarettes (SREC)

INTERVENTIONS:
Other: Nicotine patch and gum — Nicotine patch and gum will be given to subjects in the Nicotine replacement therapy cohort every visit after providing exhaled CO/Saliva cotinine test.
  Arms: counseling + nicotine replacement therapies NRT
Behavioral: Minnesota Nicotine Withdrawal Scale (MNWS) — The MNWS assesses symptoms associated with nicotine withdrawal (i.e., craving, irritability, anxiety, difficulty concentrating, restlessness, increased appetite or weight gain, depression, and insomnia).
Behavioral: ASSIST (the Alcohol, Smoking and Substance Involvement Screening) — The ASSIST is the Alcohol, Smoking and Substance Involvement Screening Test. It is a brief screening questionnaire to find out about people's use of psychoactive substances (alcohol, smoking and substance involvement).
Behavioral: Counseling — At each study visit, participants will receive counseling protocol that will be based on effective counseling manuals. The PI will train the research assistant who will assist the PI in tailoring the manual to the target group: counseling will cover health education, social support issues, and motivational enhancement to improve self-efficacy while addressing other aspects known to contribute to smoking among PLWHA (e.g., tips on dealing with depression and feeling stigmatized particularly in relation to HIV).
Other: NIDA Standardized Research E-cigarettes (SREC) — NIDA SREC has a case with a liquid tank. The e-liquid is supplied in sealed disposable cartridges that deliver >300 puffs / cartridge. The SREC uses a battery recharged via a micro USB port. A single charge is designed to outlast the capacity of an e-liquid cartridge. The e-liquid is "tobacco" flavored and contains nicotine.
  Arms: Counseling + Standardized Research E-cigarettes (SREC)

SUMMARY:
This is a research study to understand and determine the effectiveness of electronic cigarettes versus nicotine replacement therapy in adults who smoke and also live with HIV/AIDS in effort to reduce cigarette smoking.

DETAILED DESCRIPTION:
People living with HIV/AIDS (PLWHA) are known to have exceptionally higher rate of cigarette smoking and very low quit rates compared to the general population. Although a primary rationale for conducting this study is reducing health disparities among PLWHA, there is a potential benefit of the proposed work from a prevention perspective given that combustible cigarette smoking is an independent risk factor for non-adherence to ART and may decrease the effectiveness of HAART. Smoking-related illnesses are leading causes of non-HIV/AIDS-related deaths among People Living with HIV/AIDS (PLWHA). Electronic cigarettes (E-cigarettes) could help people reduce the harm of combustible cigarette (CC) through reductions in number of Cigarettes per Day (CPD) or quitting CC completely by addressing both nicotine and behavioral dependence. Unlike CC, EC are not associated with coronary heart disease or myocardial infarction. The purpose is to identify barriers and facilitators, as well as assess preliminary effectiveness of e-cigarettes as a harm reduction strategy among PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* Current Combustible Cigarette (CC) smokers (more than 5 packs in a lifetime; smokes 4 or more days/week),
* Smokes at least 10 cigarettes per day on days they smoke CC.
* Motivated to quit smoking (at least a 5 on a 10-point Likert scale).
* Must be able to provide consent
* Agree to be randomized and followed-up with,
* Reside in New York City
* Be willing to use an e-cigarette or NRT for 12 weeks.

Exclusion Criteria:

* Are pregnant (as determined by urine test) or breastfeeding (self-reported),
* State diagnosis of any medical condition (angina/heart disease) precluding use of nicotine patch or gum, or by self-report in screening questionnaire
* Reporting using NRTs or e-cigarettes or within the last 30 days
* Have untreated/are undergoing current treatment for psychiatric illness or cognitive impairment at time of initial screening as determined by the subjects' primary care doctor or a licensed study team member in screening
* Report a history of severe or untreated cardiopulmonary disease such as asthma or emphysema.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Change in Cigarettes per Day (CPD) | Visit 1 (week1), Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8), Visit 6 (week 12)
  In the e-cigarette arm, participants will be encouraged to substitute SREC (15 mg/ml nicotine in tobacco flavor) for CC in order to reduce nicotine withdrawal symptoms. Smoking reduction will be measured by a combination of self-report, text message data and changes in CO and saliva cotinine between baseline and end of treatment.

SECONDARY OUTCOMES:
Assessing differences in nicotine withdrawal symptoms | Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8)
  Will assess withdrawal symptoms of nicotine using the Minnesota Nicotine Withdrawal Scale (MNWS). The 9 item scale which assess withdrawal symptoms will be rated on a 5 point scale "not present", " slight", "mild", "moderate" and "severe" .
Assessing differences in E-cigarette dependency | Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8)
  Will assess withdrawal symptoms of E-cigarette dependency using potential side effects of NRT/SREC using the E-cigarette Dependence Index (SREC arm). 9 questions assess the experience with Electronic cigarettes to gauge how depend the subjects are on e-cigarettes (0 - 3 = not dependent, 4 - 8 low dependence, 9 - 12 medium dependence, 13+ = high dependence)
Assessing differences in nicotine use | Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8)
  Will assess withdrawal symptoms using smoking cessation self-efficacy using the Smoking Self-efficacy Questionnaire: SEQ-12. The 12 item questionnaire assess how people refrain form smoking in certain situations using a 5 point Likert scale (1=not at all sure, 2=not very sure, 3=more or less, 4=fairly sure, 5= absolutely sure).
Assessing differences in use of substance use | Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8)
  Will assess withdrawal symptoms using the acceptability through ASSIST screening tool (the Alcohol, Smoking and Substance Involvement Screening). 8 questions asking about the experience of using substances across the subjects lifetime and in the past 3 months.
Assessing differences in side effects associated with e-cigarette use | Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 6), Visit 5 (Week 8)
  Will assess withdrawal symptoms using the acceptability through self reporting questionnaire regarding demographics and tobacco use and other medications.

CONTACTS AND LOCATIONS:
Overall Officials: Omar El Shahawy, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to omar.elshahawy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.